CLINICAL TRIAL: NCT07339969
Title: The Impact of Warning Labels vs Traffic Light Labels on Food Choice and Negative Emotional Response in an Eating Disorder Population Group
Brief Title: Food Choice Among Individuals With an Eating Disorder Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Eric Robinson, Dr, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15576
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Eating Behavior Disorders
Keywords: nutrition labelling; eating disorders; food choice; warning labels; traffic light labels
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be recruited to take part in an online study where they will be required to make hypothetical food choices. Participants will complete a baseline no label task, before being randomly assigned to (1) warning label group, (2) traffic light label group, or (3) no label group in which they will complete the same task a second time (mixed design).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No label (Active Comparator): Products in the food choice task will not feature a nutrition label.
  Interventions: Behavioral: Front-of-pack nutrition labelling
- Traffic light label (Experimental): Products in the food choice task will feature a traffic light label.
  Interventions: Behavioral: Front-of-pack nutrition labelling
- Warning labels (Experimental): Products in the food choice task will feature warning labels if high in sugar, salt, fat, saturated fat, and/or calories.
  Interventions: Behavioral: Front-of-pack nutrition labelling

INTERVENTIONS:
Behavioral: Front-of-pack nutrition labelling — Participants will view a selection of six packaged food items for scenarios involving labels predominately relating to (1) sugar, (2) salt, (3) fat, (4) saturated fat, and (5) calorie content of the food products. Three items will be 'high in' that particular nutrient and three items will not be high in that nutrient. Participants will be shown all six options at once and will be asked to choose one item. In total, participants will choose five different items, one from each trial.

SUMMARY:
The aim of this study is to understand the impact of front of pack labelling systems such as, warning labels and traffic light labels on food choice and negative emotional response in an eating disorder(s) population group. Participants will be recruited to take part in an online study where they will be required to make hypothetical food choices. Participants will complete a baseline no label task, before being randomly assigned to (1) warning label group, (2) traffic light label group, or (3) no label group in which they will complete the same task a second time (mixed design). Each participant, irrespective of the group will be asked to complete five trials within the main task. Participants will view a selection of six packaged food items for scenarios involving labels predominately relating to (1) sugar, (2) salt, (3) fat, (4) saturated fat, and (5) calorie content of the food products. Three items will be 'high in' that particular nutrient and three items will not be high in that nutrient. Participants will be shown all six options at once and will be asked to choose one item. In total, participants will choose five different items, one from each trial. After participants have made their food choices for the second task, they will be asked questions about the task they have just completed.

DETAILED DESCRIPTION:
The aim of this study is to understand the impact of front of pack labelling systems such as, warning labels and traffic light labels on food choice and negative emotional response in an eating disorder(s) population group.

Hypotheses:

Both WL and TLL will affect food choice (vs. control), but WL will have a larger impact on discouraging unhealthy food choices than TLL.

Both WL and TLL will affect calorie and nutrient selected (vs. control), but WL will have a larger impact than TLL.

WL will have a larger impact on negative emotional responses than TLL.

Study type:

Randomised controlled trial (RCT).

Blinding:

Participants will not know the group to which they have been assigned to.

Additional blinding:

Participants will be given to a cover story to conceal the objectives of the study.

Study design:

Participants will be recruited to take part in an online study where they will be required to make hypothetical food choices. Participants will complete a baseline no label task, before being randomly assigned to (1) warning label group, (2) traffic light label group, or (3) no label group in which they will complete the same task a second time (mixed design).The baseline task must be completed between 24 hours and 1 week prior to completing the second task. Each participant, irrespective of the group will be asked to complete five trials within the main task. Participants will view a selection of six packaged food items for scenarios involving labels predominately relating to (1) sugar, (2) salt, (3) fat, (4) saturated fat, and (5) calorie content of the food products. Three items will be 'high in' that particular nutrient and three items will not be high in that nutrient. Participants will be shown all six options at once and will be asked to choose one item. In total, participants will choose five different items, one from each trial. After participants have made their food choices for the second task, they will be asked questions about the task they have just completed. All tasks and questionnaires will be identical in each label group - only the label will differ.

Food choice task Qualtrics XM survey software will be used to create the different trials within the food choice task. Participants will be recruited through Prolific; a data collection platform which recruits participants for online studies globally. Participants earn money by completing studies proportionate to the time it takes to complete the study (around £6 per hour). An online information sheet and consent form will be automatically displayed to participants via Qualtrics before the survey starts. Participants will be required to confirm that they have read the information sheet, and consent to taking part, in order to gain access to the survey questions. The survey will take approximately 15 minutes. Upon completion/termination of the survey, an online debrief sheet, including links to where they can be directed to for help if the study has triggered symptoms, will be automatically displayed to participants via Qualtrics.

Participants will be told to imagine they are hypothetically choosing different items for themselves to eat. The task will include 5 trials (1) crisps, (2) cereal, (3) pasta ready meal, (4) assorted savoury snacks, and (5) lunch salads. Each trial will focus on a different 'high in' nutrient, for example, (1) crisps will display 'high in salt', (2) cereals will display 'high in sugar', (3) pasta ready meals will display 'high in saturated fat', (4) assorted savoury snacks will display 'high in fat', and (5) lunch salads will display 'high in calories'. In each trial there will be three packaged food items without 'high in' labels or a 'red' traffic light label and three with WL or TLL (see "Label task questionnaire" attachment). Criteria for products labelled 'high in' is in line with labelling criteria for TLL in the UK. The design of WL will be representative of the results from patient and public involvement (PPI) from a study co-designing and examining 'high in' warning labels for a selection of food items and menu items in the UK. The design of TLL will be as it exists on UK products currently. Packaged products were selected from Tesco online supermarket. In the WL group, all TLL will be hidden. Products will be kept as similar as possible within each trial, for example, all cereals were chocolate flavoured, all crisps salt and vinegar flavoured. Pricing will not be displayed to prevent price influencing food choice.

ELIGIBILITY:
Inclusion Criteria:

* Current or past eating disorder diagnosis
* Aged 18+
* Live in the UK
* Fluent English speaker

Exclusion Criteria:

* Currently partaking in a fast or any other restrictive eating
* Any dietary restrictions/intolerances (eg. Vegan, Gluten-free, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Total number of unhealthy food items selected | Measured in both surveys, immediately after the intervention. The baseline task must be completed between 24 hours and 1 week prior to completing the second task.
  Total number of selected unhealthy food items across the 5 trials will be calculated. Unhealthy food items will be coded as items eligible for a WL or a red traffic light label for the task-specific nutrient e.g., red for salt in crisp trial.

SECONDARY OUTCOMES:
Total calories, salt, sugar, fat, saturated fat from selected food items | Measured in both surveys, immediately after the intervention.
  Total number of calories, salt (g), sugar (g), fat (g), saturated fat (g) from selected food items across the 5 trials will be calculated.
Negative emotional response | Measured in survey 2, immediately after the intervention.
  To be assessed using an adapted four-item measure, previously used to assess responses to health warning labels regarding snack selection (Clarke et al., 2020). Responses will be conveyed using seven-point scales: 'How afraid/worried/uncomfortable/disgusted does the label on food make you feel about consuming a product? With scores ranging from 1 (not at all afraid/worried/uncomfortable/disgusted) to 7 (very afraid/worried/uncomfortable/disgusted). A mean average will be calculated for the four items.
Positive and negative affect schedule (PANAS) | Measured in both surveys, pre-intervention and immediately after the intervention.
  Negative affect is to be assessed using the shortened version of PANAS (Mackinnon et al., 1999). Only the 5 items (afraid, upset, nervous, scared, distressed) that assess negative affect will be included pre and post the food choice task, as hypotheses relate to negative affect, whereas positive affect is not anticipated to be impacted by food labelling. 'How afraid/upset/nervous/scared/distressed do you feel right now?' Responses will be conveyed using Likert scale (1=Very slightly or not at all to 5= Extremely) based on the extent of which participant feels that emotion in a particular time frame (e.g., pre task and post task). Pre- and post- food choice task responses will be used to assess whether participants experience a change in negative emotion following exposure to the labels.
Reactance and avoidance | Measured in survey 2, immediately after the intervention.
  Two items will be taken from a 27-item scale developed for reactance to tobacco health warnings that were then used to assess responses to health warning labels regarding snack selection (Hall et al., 2016) (Clarke et al., 2020). Responses will be denoted using seven-point scales. Reactance: 'Are these labels annoying?'. Avoidance: 'Are you likely to avoid these labels?' With scores ranging from 1 (not annoying/not at all) to 7 (extremely annoying/very likely). Items will be scored separately.
Acceptability of labels | Measured in survey 2, immediately after the intervention.
  To be assessed using one item with responses represented on a seven point scale, adapted from a similar measure used to assess warning labels on a snack selection (Clarke et al., 2020). 'Do you support or oppose putting this label on food products?'. With scores ranging from 1 (strongly oppose) to 7 (strongly support). A score higher than the midpoint (four) will be taken as acceptability.
Perceived message effectiveness (PME) | Measured in survey 2, immediately after the intervention.
  Three items will be adapted and taken from a scale used to predict behaviour change in the context of tobacco (Baig et al., 2018). Responses will be conveyed using a Likert scale ranging from 1-5 (not at all/a great deal). Discouragement: 'This label discourages me from wanting to consume a food product'. Unpleasantness: 'The label makes consuming a food product seem unpleasant'. Concern: 'This label makes me concerned about the health effects of consuming a food product'. The mean response to the three items will be calculated.
Label awareness | Measured in survey 2, immediately after the intervention.
  'Did you notice a nutrition label when making your food choices (e.g., when choosing crisps, pasta ready meal, cereal, savoury snacks, and lunch salad?' (yes/no/unsure). If answered yes, what information was included? Response options (shown in random order): high in salt, high in sugar, high in saturated fat, high in fat, high in fibre, high in calories, calorie information, allergen information, none of these, unsure. Participants coded aware if they select all the correct responses.
Label influence | Measured in survey 2, immediately after the intervention.
  Did the presence of a nutrition label on the food items influence your food choice? Yes/No/Unsure. If answered yes, how did the nutrition label influence your food choice? Response options (shown in random order): it made me select a healthier food item, it made me avoid items high in fat/saturated fat/salt/sugar, it made me select a less healthier food item, it prompted me to think about my food choice before deciding, it didn't influence me and I ignored it, not sure.

OTHER OUTCOMES:
Aim guessing | Measured in survey 2, immediately after the intervention.
  Aim-guessing question will be included to help researchers identify whether participants are aware of the true purpose of the study. If participants correctly guess the aim, they may alter their behaviour to align with what they think the researcher expects, introducing bias. One researcher will code awareness of aims and a second researcher will independently verify the coding.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised dataset will be uploaded to the Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Indefinitely, from the date of article submission.
Access Criteria: Any interested researchers can access the anonymised dataset.